CLINICAL TRIAL: NCT07252596
Title: Pain Neuroscience Education's Effect on Memory and Pain Drawings: An Exploratory Study
Brief Title: Pain Neuroscience Education and Memory
Acronym: PNE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence In Motion (Other)
Collaborators: University of Nevada, Las Vegas (Other); Southwest Baptist University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNEMEMORY202510
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
Keywords: pain neuroscience education; Memory; Pain drawing; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a single-group assignment observational study (case series) where all participants receive the same intervention (Pain Neuroscience Education). Pre- and post-intervention measurements are taken to evaluate the effects of PNE on memory and sensory awareness in individuals with chronic pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Neuroscience Education (PNE) Intervention (Experimental): Participants will receive a standardized Pain Neuroscience Education session lasting 10 to 15 minutes, delivered by a clinician trained in advanced pain science. This educational intervention uses metaphors, examples, and images to teach patients about the biology of pain, aiming to reduce pain catastrophizing and improve cognitive and sensory outcomes.
  Interventions: Behavioral: Pain Neuroscience Education (PNE)

INTERVENTIONS:
Behavioral: Pain Neuroscience Education (PNE) — A 10-15 minute individualized educational session focusing on the neuroscience of pain. The session aims to reconceptualize the patient's understanding of their chronic pain by explaining the underlying biological, cognitive, and emotional mechanisms involved. Clinicians use a standardized checklist of metaphors and teaching tools tailored to the patient's clinical presentation.

SUMMARY:
Brief Summary:

The goal of this observational study (case series) is to determine whether Pain Neuroscience Education (PNE) can influence memory function and sensory awareness in adults (18 years and older) experiencing chronic pain lasting more than one year.

The main questions it aims to answer are:

Does a single PNE session improve memory performance, as measured by the Montreal Cognitive Assessment (MoCA)?

Does PNE change sensory awareness, as represented by alterations in body pain drawings using a grid overlay method?

Participants will:

Complete pre-intervention assessments, including:

Numeric Pain Rating Scale (NPRS)

Body chart drawing to map pain area

Montreal Cognitive Assessment (MoCA)

Pain Catastrophization Scale (PCS)

Receive a 10-15 minute standardized PNE session delivered by a licensed clinician trained in pain science

Complete the same assessments immediately after the intervention to identify any changes in memory, sensory awareness, and pain perception

This study aims to explore whether PNE can positively impact cognitive and sensory functions affected by chronic pain, beyond its already-established effects on movement and pain intensity.

DETAILED DESCRIPTION:
Detailed Description:

Chronic pain is a complex, multidimensional condition affecting approximately 25% of the global population. It is increasingly understood through the lens of brain-based changes, particularly the dynamic pain connectome, a network of brain regions involved in sensory, cognitive, and emotional processing. Functional reorganization in chronic pain patients may contribute to clinical symptoms beyond pain, such as memory loss, decreased sensory awareness, and altered motor control.

Pain Neuroscience Education (PNE) is an educational intervention that aims to reconceptualize a patient's understanding of pain to reduce fear-avoidance, pain catastrophization, and disability. Systematic reviews have demonstrated its effectiveness in reducing pain and improving movement. Early fMRI studies suggest that PNE may also deactivate pain-related brain areas and normalize brain function.

This case series seeks to explore the impact of a single PNE session on cognitive (memory) and sensory (body perception) outcomes in individuals with chronic pain. Participants (aged 18 and older) who meet inclusion criteria and consent to the study will undergo pre- and post-intervention assessments. These include:

Numeric Pain Rating Scale (NPRS)

Pain body chart (grid overlay method)

Montreal Cognitive Assessment (MoCA)

Pain Catastrophization Scale (PCS)

Following baseline assessments, participants will receive a 10-15 minute individualized PNE session delivered by licensed clinicians trained in advanced pain science. Immediately post-intervention, assessments will be repeated to evaluate changes.

The study aims to contribute to the understanding of how PNE may influence brain-related symptoms associated with chronic pain, specifically memory function and sensory mapping. Findings could provide early evidence to support broader applications of PNE beyond movement-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Chronic pain > 1 year
* Provide written consent
* Proficient in reading and understanding English

Exclusion Criteria:

* Not willing to participate in the study
* Have received PNE as a treatment before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Memory Function (Montreal Cognitive Assessment - MoCA) | At baseline (prior to the pain neuroscience education session) and immediately after completion of the treatment session
  Description: Change in MoCA score to assess improvement or decline in cognitive function, particularly memory, associated with chronic pain. The MoCA is scored out of 30; a change of 2 points or more is considered clinically meaningful.
Sensory Awareness (Body Chart Pain Area - Grid Overlay Count) | At baseline (prior to the pain neuroscience education session) and immediately after completion of the treatment session
  Change in the number of grid blocks marked on the body pain chart to quantify alteration in perceived pain area, reflecting somatosensory representation changes.

SECONDARY OUTCOMES:
Self-Reported Pain Intensity (Numeric Pain Rating Scale - NPRS) | At baseline (prior to the pain neuroscience education session) and immediately after completion of the treatment session
  Change in pain intensity reported by the patient on an 11-point scale (0-10). The minimal clinically important difference (MCID) is 1.7 points.
Pain Catastrophization (Pain Catastrophization Scale - PCS) | At baseline (prior to the pain neuroscience education session) and immediately after completion of the treatment session
  Change in PCS scores assessing catastrophic thinking related to pain on a 13-item, 5-point Likert scale. Higher scores indicate greater catastrophizing.

OTHER OUTCOMES:
Demographic and Clinical Characteristics | Baseline, pre-intervention
  Age, gender, ethnicity, pain location, pain duration, family history of pain, presence of memory loss, and spreading of pain since onset.
Clinician Checklist | Immediately after intervention
  Clinician-reported pain phenotype, diagnosis, metaphors used during PNE, and rating of therapeutic alliance to explore potential influences on intervention effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Louw, PT, PhD, Principal Investigator — Evidence In Motion

IPD SHARING:
Plan to Share IPD: No
Sharing IPD requires time, personnel, infrastructure, and data curation, which might not be feasible due to funding or staffing limitations. In addition, the informed consent documents do not include a provision for IPD sharing.
  Participants have not agreed to data sharing beyond the original study purpose.

REFERENCES:
- [Background] Sullivan MJL, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment
- [Background] Lansdall CJ, McDougall F, Butler LM, Delmar P, Pross N, Qin S, McLeod L, Zhou X, Kerchner GA, Doody RS. Establishing Clinically Meaningful Change on Outcome Assessments Frequently Used in Trials of Mild Cognitive Impairment Due to Alzheimer's Disease. J Prev Alzheimers Dis. 2023;10(1):9-18. doi: 10.14283/jpad.2022.102. PMID 36641605
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Sanders NW, Mann NH 3rd, Spengler DM. Pain drawing scoring is not improved by inclusion of patient-reported pain sensation. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2735-41; discussion 2742-3. doi: 10.1097/01.brs.0000244674.99258.f9. PMID 17077744
- [Background] Lacey RJ, Lewis M, Jordan K, Jinks C, Sim J. Interrater reliability of scoring of pain drawings in a self-report health survey. Spine (Phila Pa 1976). 2005 Aug 15;30(16):E455-8. doi: 10.1097/01.brs.0000174274.38485.ee. PMID 16103839
- [Background] Matthews M, Rathleff MS, Vicenzino B, Boudreau SA. Capturing patient-reported area of knee pain: a concurrent validity study using digital technology in patients with patellofemoral pain. PeerJ. 2018 Mar 8;6:e4406. doi: 10.7717/peerj.4406. eCollection 2018. PMID 29568700
- [Background] Wand BM, Keeves J, Bourgoin C, George PJ, Smith AJ, O'Connell NE, Moseley GL. Mislocalization of sensory information in people with chronic low back pain: a preliminary investigation. Clin J Pain. 2013 Aug;29(8):737-43. doi: 10.1097/AJP.0b013e318274b320. PMID 23835768
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Kregel J, Meeus M, Malfliet A, Dolphens M, Danneels L, Nijs J, Cagnie B. Structural and functional brain abnormalities in chronic low back pain: A systematic review. Semin Arthritis Rheum. 2015 Oct;45(2):229-37. doi: 10.1016/j.semarthrit.2015.05.002. Epub 2015 May 16. PMID 26092329
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] Suso-Marti L, Cuenca-Martinez F, Alba-Quesada P, Munoz-Alarcos V, Herranz-Gomez A, Varangot-Reille C, Dominguez-Navarro F, Casana J. Effectiveness of Pain Neuroscience Education in Patients with Fibromyalgia: A Systematic Review and Meta-Analysis. Pain Med. 2022 Oct 29;23(11):1837-1850. doi: 10.1093/pm/pnac077. PMID 35587171
- [Background] Krebs-Roubicek E, Osterwalder R. [Gerontopsychiatry--collaboration between inpatient and outpatient care]. Ther Umsch. 1986 Jan;43(1):69-74. No abstract available. German. PMID 3952688
- [Background] Rastegarnia S, St-Laurent M, DuPre E, Pinsard B, Bellec P. Brain decoding of the Human Connectome Project tasks in a dense individual fMRI dataset. Neuroimage. 2023 Dec 1;283:120395. doi: 10.1016/j.neuroimage.2023.120395. Epub 2023 Oct 12. PMID 37832707
- [Background] Smallwood RF, Laird AR, Ramage AE, Parkinson AL, Lewis J, Clauw DJ, Williams DA, Schmidt-Wilcke T, Farrell MJ, Eickhoff SB, Robin DA. Structural brain anomalies and chronic pain: a quantitative meta-analysis of gray matter volume. J Pain. 2013 Jul;14(7):663-75. doi: 10.1016/j.jpain.2013.03.001. Epub 2013 May 17. PMID 23685185
- [Background] Hashmi JA, Baliki MN, Huang L, Baria AT, Torbey S, Hermann KM, Schnitzer TJ, Apkarian AV. Shape shifting pain: chronification of back pain shifts brain representation from nociceptive to emotional circuits. Brain. 2013 Sep;136(Pt 9):2751-68. doi: 10.1093/brain/awt211. PMID 23983029
- [Background] Moseley GL. Evidence for a direct relationship between cognitive and physical change during an education intervention in people with chronic low back pain. Eur J Pain. 2004 Feb;8(1):39-45. doi: 10.1016/S1090-3801(03)00063-6. PMID 14690673
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Liao WW, Wu CY, Liu CH, Lin SH, Chiau HY, Chen CL. Test-retest reliability and minimal detectable change of the Contextual Memory Test in older adults with and without mild cognitive impairment. PLoS One. 2020 Jul 31;15(7):e0236654. doi: 10.1371/journal.pone.0236654. eCollection 2020. PMID 32735628
- [Background] Gerhardt A, Eich W, Janke S, Leisner S, Treede RD, Tesarz J. Chronic Widespread Back Pain is Distinct From Chronic Local Back Pain: Evidence From Quantitative Sensory Testing, Pain Drawings, and Psychometrics. Clin J Pain. 2016 Jul;32(7):568-79. doi: 10.1097/AJP.0000000000000300. PMID 26379077
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Siddall B, Ram A, Jones MD, Booth J, Perriman D, Summers SJ. Short-term impact of combining pain neuroscience education with exercise for chronic musculoskeletal pain: a systematic review and meta-analysis. Pain. 2022 Jan 1;163(1):e20-e30. doi: 10.1097/j.pain.0000000000002308. PMID 33863860
- [Background] Wood L, Hendrick PA. A systematic review and meta-analysis of pain neuroscience education for chronic low back pain: Short-and long-term outcomes of pain and disability. Eur J Pain. 2019 Feb;23(2):234-249. doi: 10.1002/ejp.1314. Epub 2018 Oct 14. PMID 30178503
- [Background] Kucyi A, Davis KD. The dynamic pain connectome. Trends Neurosci. 2015 Feb;38(2):86-95. doi: 10.1016/j.tins.2014.11.006. Epub 2014 Dec 22. PMID 25541287
- [Background] Moseley GL. Widespread brain activity during an abdominal task markedly reduced after pain physiology education: fMRI evaluation of a single patient with chronic low back pain. Aust J Physiother. 2005;51(1):49-52. doi: 10.1016/s0004-9514(05)70053-2. PMID 15748125
- [Background] Louw A, Puentedura EJ, Diener I, Peoples RR. Preoperative therapeutic neuroscience education for lumbar radiculopathy: a single-case fMRI report. Physiother Theory Pract. 2015;31(7):496-508. doi: 10.3109/09593985.2015.1038374. PMID 26395827
- [Background] Puentedura EJ, Louw A. A neuroscience approach to managing athletes with low back pain. Phys Ther Sport. 2012 Aug;13(3):123-33. doi: 10.1016/j.ptsp.2011.12.001. Epub 2011 Dec 27. PMID 22814445
- [Background] Melzack R. Pain and the neuromatrix in the brain. J Dent Educ. 2001 Dec;65(12):1378-82. PMID 11780656
- [Background] Moseley GL. A pain neuromatrix approach to patients with chronic pain. Man Ther. 2003 Aug;8(3):130-40. doi: 10.1016/s1356-689x(03)00051-1. PMID 12909433
- [Background] Nahin RL, Feinberg T, Kapos FP, Terman GW. Estimated Rates of Incident and Persistent Chronic Pain Among US Adults, 2019-2020. JAMA Netw Open. 2023 May 1;6(5):e2313563. doi: 10.1001/jamanetworkopen.2023.13563. PMID 37191961
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Moseley GL. Reconceptualising pain acording to modern pain sciences. Physical Therapy Reviews. 2007;12:169-178.
- [Background] Zimney K, Van Bogaert W, Louw A. The Biology of Chronic Pain and Its Implications for Pain Neuroscience Education: State of the Art. J Clin Med. 2023 Jun 21;12(13):4199. doi: 10.3390/jcm12134199. PMID 37445234
- [Background] George SZ, Valencia C, Beneciuk JM. A psychometric investigation of fear-avoidance model measures in patients with chronic low back pain. J Orthop Sports Phys Ther. 2010 Apr;40(4):197-205. doi: 10.2519/jospt.2010.3298. PMID 20357418